CLINICAL TRIAL: NCT06070948
Title: A Bioavailability and Food Effect Study of Venetoclax New High Drug Load Tablet Formulation in Healthy Female Subjects
Brief Title: A Study to Assess Food Effect of Venetoclax New Tablet Formulation in Healthy Female Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M22-457
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers
Keywords: Venetoclax
MeSH Terms: interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Regimen A (Experimental): Participants will receive venetoclax dose A commercial formulation following a high-fat meal.
  Interventions: Drug: Venetoclax
- Regimen B (Experimental): Participants will receive venetoclax dose B new formulation following a high-fat meal.
  Interventions: Drug: Venetoclax
- Regimen C (Experimental): Participants will receive venetoclax dose A new formulation following a high-fat meal.
  Interventions: Drug: Venetoclax
- Regimen D (Experimental): Participants will receive venetoclax dose B new formulation under fasted conditions.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Oral; Tablet

SUMMARY:
The purpose of this study is to assess the bioavailability of two different doses of venetoclax new high drug load formulation tablets relative to two tablets of the currently marketed venetoclax tablets under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is >= 18.0 to <= 32.0 kg/m2 after rounding to the tenths decimal.
* A condition of general good health based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
* Participant must be postmenopausal, permanently surgically sterile, or perimenopausal or premenopausal and practicing a method of birth control until at least 1 month after the last dose of study drug.

Exclusion Criteria:

- History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Venetoclax | Up to Day 27
  Cmax of Venetoclax will be assessed.
Time to Cmax (Tmax) of Venetoclax | Up to Day 27
  Tmax of Venetoclax will be assessed.
Area Under the Plasma Concentration-time Curve (AUC) from Time 0 to the Last Measurable Concentration (AUCt) of Venetoclax | Up to Day 27
  AUCt of Venetoclax will be assessed.
AUC from Time 0 to Infinity (AUCinf) of Venetoclax | Up to Day 27
  AUCinf of Venetoclax will be assessed.
Apparent Terminal Phase Elimination Rate Constant (β, BETA) of Venetoclax | Up to Day 27
  Apparent terminal phase elimination rate constant (β, BETA) of Venetoclax will be assessed.
Terminal Phase Elimination Half-life (t1/2) of Venetoclax | Up to Day 27
  Terminal phase elimination half-life (t1/2) of Venetoclax will be assessed.
Number of Adverse Events (AEs) | Baseline to Day 57
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 259897, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-457